CLINICAL TRIAL: NCT01643278
Title: Phase I Study of Dasatinib in Combination With Ipilimumab for Patients With Advanced Gastrointestinal Stromal Tumor and Other Sarcomas
Brief Title: Dasatinib and Ipilimumab in Treating Patients With Gastrointestinal Stromal Tumors or Other Sarcomas That Cannot Be Removed by Surgery or Are Metastatic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01165; NCI-2012-01165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000737378; 12-083; 9172 (Other: Memorial Sloan-Kettering Cancer Center); 9172 (Other: CTEP); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Gastrointestinal Stromal Tumor; Stage III Soft Tissue Sarcoma; Stage IV Soft Tissue Sarcoma
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma | interventions — Dasatinib; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (dasatinib and ipilimumab) (Experimental): Patients receive dasatinib PO QD for 7 days. Patients then receive dasatinib PO QD and ipilimumab IV once on weeks 1, 4, 7 and 10. Beginning on week 24, patients then receive dasatinib PO QD and ipilimumab IV once every 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of dasatinib when given together with ipilimumab in treating patients with gastrointestinal stromal tumors or other sarcomas that cannot be removed by surgery or have spread to other places in the body. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as ipilimumab, can block tumor growth in different ways by targeting certain cells. Giving dasatinib together with ipilimumab may be a better treatment for patients with gastrointestinal stromal tumors or other sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of treatment with ipilimumab in combination with dasatinib in subjects with gastrointestinal stromal tumor (GIST) and other advanced sarcomas.

SECONDARY OBJECTIVES:

I. Response rate (RR) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, immune-related response criteria, and Choi criteria.

II. Progression free survival (PFS). III. Progression-free survival at 6 months (PFS6months). IV. Overall survival (OS). V. Immunological correlative studies.

OUTLINE: This is a dose-escalation study of dasatinib.

Patients receive dasatinib orally (PO) once daily (QD) for 7 days. Patients then receive dasatinib PO QD and ipilimumab intravenously (IV) once on weeks 1, 4, 7 and 10. Beginning on week 24, patients then receive dasatinib PO QD and ipilimumab IV once every 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* DOSE ESCALATION COHORT: subjects must have histologically or cytologically confirmed sarcoma that is metastatic or unresectable
* DOSE EXPANSION COHORT: subjects must have histologically or cytologically confirmed GIST that is metastatic or unresectable
* Patients must have measurable disease per RECIST 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* DOSE ESCALATION COHORT: patients must have had at least one prior therapy
* DOSE EXPANSION COHORT: GIST patients must have had progression on or have been intolerant to imatinib and sunitinib
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3 K/mcL
* Absolute neutrophil count >= 1.5 K/mcL
* Platelets >= 100 K/mcL
* Hemoglobin >= 8.0 g/dl
* Total bilirubin =< 1.5 x institutional upper limit of normal; note: patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the treating physician and/or the principal investigator
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of dasatinib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy (non-tyrosine kinase inhibitor [TKI]) or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients with a history of prior treatment with ipilimumab or dasatinib
* Patients who are receiving any other investigational agents
* Patients with known brain metastases are excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to dasatinib and ipilimumab
* Patients who require concurrent treatment with any medications or substances that are potent inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)
* Patients who require concurrent treatment with any medications or substances that have significant proarrhythmic potential are ineligible
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain dasatinib tablets are excluded
* Patients may not have any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged corrected QT interval (QTc) > 480 msec
  * Ejection fraction less than 50%
  * Major conduction abnormality (unless a cardiac pacemaker is present)
* Uncontrolled intercurrent illness including, but not limited to, the following: ongoing or active infection; history of significant bleeding disorder, including congenital (von Willebrand's disease) or acquired (anti-factor VIII antibodies) disorders; large pleural effusions; or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with dasatinib
* Subjects may not have known human immunodeficiency virus (HIV), active hepatitis A, or hepatitis B or C infection
* Subjects with any active autoimmune disease or a documented history of autoimmune disease or history of syndrome that required systemic steroids or immunosuppressive medications including but not limited to inflammatory bowel disease, rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (e.g. Guillain-Barre syndrome), and multiple sclerosis; patients with vitiligo, asthma and diabetes are NOT excluded; final determination can be left to the discretion of the principal investigator
* Subjects may not have ongoing chronic diarrhea
* Subjects may not have had prior organ allograft or allogeneic bone marrow transplantation
* Subjects may not have any major surgery within 4 weeks
* Subjects may not have known current drug or alcohol abuse
* Subjects may not have an underlying medical condition that in the opinion of the investigator could adversely affect the ability of the subject to comply with or tolerate study procedures and/or study therapy, or confound the ability to interpret the tolerability of combined administration of dasatinib and ipilimumab in treated subjects
* Subjects may not have other active malignancies other than indolent malignancies not requiring active therapy which the investigator determines are unlikely to interfere with treatment and safety analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the highest dose studied for which the observed incidence of dose-limiting toxicity is less than 33% according to the National Cancer Institute Common Toxicity Criteria | Up to week 12
  Frequencies of toxicities will be tabulated.

SECONDARY OUTCOMES:
OS as measured by RECIST 1.1, Choi and immune-related response criteria | Up to 3 years
  Will be estimated using Kaplan-Meier methodology.
PFS as measured by RECIST 1.1, Choi and immune-related response criteria | From start of treatment to time of progression or death, whichever occurs first, assessed up to 3 years
  Will be estimated using Kaplan-Meier methodology.
PFS at 6 months as measured by RECIST 1.1, Choi and immune-related response criteria | 6 months
  Will be estimated using Kaplan-Meier methodology.
RR as measured by RECIST 1.1, Choi and immune-related response criteria | Up to 3 years
  Immune related response rate (complete response + partial response) and Choi criteria will be calculated along with a 95% confidence interval.

OTHER OUTCOMES:
Change in humoral and cellular immune response | Baseline to up to 4 weeks after treatment
  Relationships between clinical response, lymphocyte phenotype, cytokines, and effect of dasatinib and ipilimumab on humoral and cellular immune responses will be evaluated. Summary statistics for peripheral blood biomarkers of immunoregulatory activity (T-cell subpopulation counts, cytokines, and corresponding changes [or % changes]) will be tabulated by study day/dose. Time courses of biomarker measures will be investigated graphically; further analysis may be performed to characterize relationships. Associations between changes and dasatinib exposure will be explored graphically.
Change in tumor immunological markers in patients treated at the expansion cohort (as of May 2015 patients on expansion cohort will not undergo protocol biopsies) | Baseline to up to week 6
  Summary statistics for measures and changes from baseline of tumor-based markers including T-cell (cluster of differentiation [CD] 4, CD8, CD45, forkhead box P3), apoptosis markers, and indoleamine 2,3-dioxygenase 1/2 will be tabulated. Associations between biomarkers and efficacy measures will be analyzed in all response-evaluable subjects.
Downstream molecular effects of therapy on tumor viability as measured by changes in KIT expression and secondary mutations in resistant tumor specimens | Baseline to up to 4 weeks after treatment
  Changes will be correlated with tumor response by Fisher's exact test.
Genotype (v-Kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog [KIT] and platelet-derived growth factor receptor-alpha [PDGFR-a]) mutation status | Baseline
  Associations of mutation status with response rate and PFS6months will be assessed using Fisher's exact test. Associations of mutation status with PFS and overall survival will be assessed using the log rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D'Angelo, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States